06/03/2025 v1.1

IRAS ID: 341922



IRAS ID: 341922

Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project: A study to explore the feasibility and efficacy of Group Traumatic Episode Protocol (GTEP) for reducing trauma symptoms in individuals following a traumatic birthing experience.

individuals following a traumatic birthing experience. Name of Researcher: Grace Rodgers Please initial box I confirm that I have read the participant information sheet (version 1.1, dated 06/03/2025) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. I understand that should I withdraw before the study has finished, any data already collected may be used in data analysis. I understand the research team will arrange a home visit to confirm my eligibility for the study and if I am eligible I 3. will start the study. 4. I understand that relevant sections of my medical records and data collected during the study, may be looked at by individuals from the sponsor, regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to access my records. 5. I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers. I agree to my General Practitioner being informed of my participation in the study. This may include any necessary exchange of information about me between my GP and the research team, should there be any concerns about safety. 7. I understand that the data held on my clinical records will be accessed by the research team to provide information for the study (e.g., demographic information including age and ethnicity, contact details). I understand that my anonymised data will be used for dissemination in publications (e.g., within scientific journals/conference abstracts). This might include anonymised quotes. I agree to take part in the above study. 9.

06/03/2025 v1.1

IRAS ID: 341922



| Name of Participant | Date | Signature |
|---|---|---|
| Name of Person | Date | Signature |
| seeking consent | | |
| For verbal witnessed co | nsent only: | |
| Name of Witness | Date | Signature |
| (OPTIONAL) If you wou | ld like to receive the results of the | s study when it is complete, please provide your email address below: |
| (OPTIONAL) If you would like to receive the results of the study when it is complete, please provide your email address below: | | |